CLINICAL TRIAL: NCT05997771
Title: A Personal Nutrition Advisor to Assist Remote Dietary Counselling for Weight Loss and Maintenance
Acronym: PNA-ORIGINATE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lia Bally (Other)
Responsible Party: Sponsor-Investigator, Lia Bally, Prof. Dr.med. et Dr. phil., Insel Gruppe AG, University Hospital Bern
Organization: Insel Gruppe AG, University Hospital Bern (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: PNA-ORIGINATE
Record Dates: First submitted 2023-06-15; First posted 2023-08-18 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-06

CONDITIONS: Obesity
Keywords: Nutritional counselling; Personalised nutrition; Dietary advice; Usability
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Intervention Model Description: The evaluation of the usability will be done using a prospective single arm design (n=80). In addition, we will collect data regarding the efficacy of the intervention by comparing results of the study participants to results of historical controls (n=80). Historical controls are patients receiving the same usual care dietary counselling as the study participants but without assistance by the personal nutrition advisor.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study Intervention Group (Experimental): The study intervention group will be undergoing 3 months of Personalized Nutrition Advisor (PNA)-assisted remote nutritional counselling.The PNA data analysis tool will be used by the dietitians during remote nutritional counselling sessions.The service will be delivered to patients undergoing GLP-1 based obesity treatment as part of their usual care. The study intervention group will report treatment-satisfaction and self-efficacy via questionnaires at baseline, 1.5 - and 3 months.
  Patients who expressed their interest in participating in a focus group at the time of study inclusion, will be invited for a 60 min online interview session chaired by an experienced moderator. The focus group will consists of a maximum of 10 participants and address the patient's perspective on the utility of the dietitians' advice, discrepancy from expectations, general feedback and suggestions for PNA improvement using a semi structured discussion guide held in an open and spontaneous format
  Interventions: Other: Personal Nutrition Advisor

INTERVENTIONS:
Other: Personal Nutrition Advisor — The study intervention will be the use of the PNA data analysis tool during remote nutritional counselling sessions delivered by certified dietitians, also referred to as PNA-assisted remote nutritional counselling.

SUMMARY:
The purpose of the study is to assess the usability of the PNA and satisfaction with the treatment within the framework of usual care remote nutritional counselling for GLP-1-supported weight management and collect pilot data on its potential to support weight loss.

DETAILED DESCRIPTION:
The global prevalence of obesity and overweight is increasing and persistently drives global mortality and morbidity.As overweight and obesity are the result of an imbalance between energy intake and energy use, achieving a negative energy balance build the foundation for weight loss. Whilst dietary modification as a standalone procedure often fail in achieving or maintaining weight loss, the recent advent of supportive Glucagon-like Peptide-1 (GLP-1) based pharmacotherapies have greatly changed the landscape.Dietary counselling help people on GLP-1 based treatment reaching their individual weight goals and continued reimbursement of medication costs. However, nutritional advice provided by dietitians is often generic, not sufficiently aligned to individual weight loss trajectories.

The "Personal Nutrition Advisor" (PNA) is a decision support tool which is built upon an interpretable weight prediction model based on the energy balance equation (energy intake is a function of recorded dietary intake and a latent part dependent on observed weight changes, whereas energy expenditure is a function of weight and physical activity). Food, weight- and activity records captured using a smartphone application represent input data to the model. Output of the model is the predicted body weight trajectory alongside with personalized recommendations to reach a pre-defined target weight.

Integrating the PNA into a remote dietary counselling programme, in which certified dietitians deliver nutritional and lifestyle coaching via an application, has the potential to improve treatment satisfaction and efficacy. Therefore, the purpose of the study assess the usability of the PNA and satisfaction with the treatment within the framework of usual care remote nutritional counselling for GLP-1-supported weight management and collect pilot data on its potential to support weight loss.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Receiving GLP-1-based pharmacotherapy in combination with remote nutritional counselling
* Achieved weight loss of ≥5 (for baseline BMI 28-35 kg/m2) or ≥7% (for baseline BMI≥35kg/m2) after 4 months of GLP-1 based therapy (1st milestone)

Exclusion Criteria:

* Inability to give written informed consent
* Any physical or psychological disease or condition likely to interfere with the normal conduct of the study and interpretation of the study results
* Self-reported pregnancy, planed pregnancy within next 3 months or breast-feeding
* Concomitant participation in another trial that interferes with the normal conduct of the study and interpretation of the study results
* Not proficient in German

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2023-08-25 (Actual); Primary Completion 2024-04-22 (Actual); Study Completion 2024-05-06 (Actual)

PRIMARY OUTCOMES:
Change in the overall mean satisfaction score of the Nutritional and Dietetic Patient Outcomes Questionnaire (NDPOQ) | From baseline to 3 months of the respective study period
  This outcome will evaluate the patient treatment satisfaction with the counselling of the "Personal Nutrition Advisor" (PNA) -assisted remote nutritional counselling. The NDPOQ includes a 5 point likert scale of agreement (5 points=strongly agree, 1 point= strongly disagree) of 15 questions.
The overall mean score of the "perceived impact" section from the user version of the mobile application scale (uMARS ) | Post intervention visit (3 months after baseline)
  This outcome will evaluate patient satisfaction with the counselling of the "Personal Nutrition Advisor" (PNA) -assisted remote nutritional counselling. The uMARS includes a 5 point likert scale of agreement (5 points=strongly agree, 1 point= strongly disagree) of 5 questions.
The overall mean score of the Healthcare Systems Usability Scale (HSUS) | Post intervention visit (3 months after baseline)
  This outcome will evaluate dietitian reported usability of the "Personal Nutrition Advisor" (PNA)- assisted remote nutritional counselling. HSUS includes a 5 point likert scale of agreement (5 points=strongly agree, 1 point= strongly disagree) of 20 questions.

SECONDARY OUTCOMES:
Change in self reported weight (%) | From baseline to 3 months of the respective study period
  This outcome will evaluate the potential to support weight loss by PNA-assisted remote nutritional counselling (self-reported weight closest to start and end of the study period).
Proportion of patients reaching >5% weight loss | At start of the GLP-1 based pharmacotherapy to 3 months of the respective study period
  This outcome will evaluate the potential to support weight loss by PNA-assisted remote nutritional counselling (calculated from the initial weight, measured in-clinic at start of the GLP-1 based pharmacotherapy)
Proportion of patients reaching >10% weight loss | At start of the GLP-1 based pharmacotherapy to 3 months of the respective study period
  This outcome will evaluate the potential to support weight loss by PNA-assisted remote nutritional counselling (calculated from the initial weight, measured in-clinic at start of the GLP-1 based pharmacotherapy)
Proportion of patients reaching >15% weight loss | At start of the GLP-1 based pharmacotherapy to 3 months of the respective study period
  This outcome will evaluate the potential to support weight loss by PNA-assisted remote nutritional counselling (calculated from the initial weight, measured in-clinic at start of the GLP-1 based pharmacotherapy)
Change in daily number of logged meals and beverages | From the first day of the respective study period to 3 months thereafter
  This outcome will evaluate the impact of PNA-assisted remote nutritional counselling on frequency of dietary self-monitoring (manual entries of pictures, text tags and food/beverage tags per day)
Change in energy intake (kcal/day) | From the first day of the respective study period to 3 months thereafter
  This outcome will evaluate the impact of PNA-assisted remote nutritional counselling on PNA derived dietary intake, calculated by the energy balance model embedded in the PNA using manual entries of weight logs, meal logs and activity logs.
Change in energy expenditure (kcal/day) | From the first day of the respective study period to 3 months thereafter
  This outcome will evaluate the impact of PNA-assisted remote nutritional counselling on PNA derived dietary expenditure, calculated by the energy balance model embedded in the PNA using manual entries of weight logs, meal logs and activity logs.
Change in relative carbohydrate content (%) | From the first day of the respective study period to 3 months thereafter
  This outcome will evaluate the impact of PNA-assisted remote nutritional counselling on PNA derived nutrient distribution, calculated by the energy balance model embedded in the PNA using manual entries of weight logs, meal logs and activity logs.
Change in relative protein content (%) | From the first day of the respective study period to 3 months thereafter
  This outcome will evaluate the impact of PNA-assisted remote nutritional counselling on PNA derived nutrient distribution, calculated by the energy balance model embedded in the PNA using manual entries of weight logs, meal logs and activity logs.
Change in relative fat content (%) | From the first day of the respective study period to 3 months thereafter
  This outcome will evaluate the impact of PNA-assisted remote nutritional counselling on PNA derived nutrient distribution, calculated by the energy balance model embedded in the PNA using manual entries of weight logs, meal logs and activity logs.
Change in relative fiber content (%) | From the first day of the respective study period to 3 months thereafter
  This outcome will evaluate the impact of PNA-assisted remote nutritional counselling on PNA derived nutrient distribution, calculated by the energy balance model embedded in the PNA using manual entries of weight logs, meal logs and activity logs.
Change in self-reported exercise engagement per week (hours/week) | At baseline and at 3 months of study intervention
  This outcome will evaluate the impact of PNA-assisted remote nutritional counselling on self-reported physical activity using manual entries of activity logs.
Change in the overall mean score of the General Self-efficacy Scale (GSE) from Imperial College London | From baseline to 3 months of the respective study period
  This outcome will evaluate the impact of PNA-assisted remote nutritional counselling on self-efficacy. GSE includes a 5 point Likert scale of confidence (Not at all confident =1 point, Extremely confident=5 points) of 6 questions.
Collection of open ended PNA specific feedback questionnaires | Post intervention visit (3 months after baseline)
  This qualitative outcome will collect opinions from patients and dietitians regarding the components of the PNA with the aim to further optimise its perceived usefulness.
Qualitative collection of patient reported PNA specific feedback. | Post intervention visit (3 months after baseline)
  This qualitative outcome will be assessed by an semi structured remote patient group interview addressing the patient's perspective on the utility of the dietitians' advice, discrepancy from expectations, general feedback and suggestions for PNA improvement.

CONTACTS AND LOCATIONS:
Overall Officials: Lia Bally, MD-PhD, Principal Investigator — Inselspital University Hospital Bern, University of Bern
Locations (1):
- Department of Diabetes, Endocrinology, Clinical Nutrition and Metabolism, Inselspital, Bern University Hospital, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
Anonymised individual participant data will be shared after inquiry via a validated sharing platform (yet to be defined). Anonymised data packages will be available once the final study results are published in a peer-reviewed journal.
Supporting Information: Study Protocol
Time Frame: After publication of the study results in a peer-reviewed journal
Access Criteria: Contact with an approval by the corresponding author